CLINICAL TRIAL: NCT04510363
Title: Optic Nerve Sheath Diameter, Carotid Duplex and Transcranial Duplex as a Prognostic Predicting Factor in Post-cardiac Arrest Patients
Brief Title: Optic Nerve Sheath Diameter, Carotid Duplex and Transcranial Duplex as a Prognostic Factor
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201911027RINC
Record Dates: First submitted 2020-08-02; First posted 2020-08-12 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Neurologic Dysfunction
MeSH Terms: conditions — Neurologic Manifestations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (2):
- cardiac arrest survivors: cardiac arrest survivors
- age- and sex-matched controls: age- and sex-matched controls

SUMMARY:
Optic nerve sheath diameter (ONSD) had been proved to be associated with increased intracranial pressure and can be used as one of the prognostic factors in cardiac arrest patients. It is simple, quick and can be measured repeatedly. Carotid duplex and transcranial duplex(TCD) provide rapid, noninvasive, real-time measures of cerebrovascular function. It can be used to assess the vascular territory by measuring blood flow, and to evaluate factors include brain perfusion, plaque morphology, and patency of intracranial collaterals. Hence, it could act as a crucial role in neuroprognosis in post-arrest patients. In this study, the investigator aimed to analyze the ONSD diameters, ONSD/external transverse diameter (ETD) ratio, carotid duplex and transcaranial duplex parameters in different stages of post-cardiac arrest care, demographic characteristics and resuscitation information with the neurological outcome of post-cardiac arrest patients. The ONSD diameter, and ONSD/ETD ratio were compared with age-, and sex-matched normal volunteers.

DETAILED DESCRIPTION:
Prediction of the neurological outcome in resuscitated post-cardiac arrest patients is important to tailor appropriate management plans. Brain imaging, electrophysiological evaluations, biomarkers all take part in neuroprognosis in cardiac arrest patients, however, these modalities are more expensive or not suitable to repeat in a short time. Optic nerve sheath diameter (ONSD) had been proved to be associated with increased intracranial pressure2 and can be used as one of the prognostic factors in cardiac arrest patients. It is simple, quick and can be measured repeatedly. Carotid duplex and transcranial duplex(TCD) provide rapid, noninvasive, real-time measures of cerebrovascular function. It can be used to assess the vascular territory by measuring blood flow, and to evaluate factors include brain perfusion, plaque morphology, and patency of intracranial collaterals.

Hence, it could act as a crucial role in neuroprognosis in post-arrest patients. In this study, the investigator aimed to analyze the ONSD diameters, ONSD/ETD ratio, carotid duplex and transcaranial duplex parameters in different stages of post-cardiac arrest care, demographic characteristics and resuscitation information with the neurological outcome of post-cardiac arrest patients.

ELIGIBILITY:
Inclusion Criteria:

. Non-traumatic cardiac arrest adult patients achieving return of spontaneous circulation after resuscitation

Exclusion Criteria:

* traumatic cardiac arrests
* non-traumatic arrest patients without return of spontaneous circulation after resuscitation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-traumatic cardiac arrest adult patients achieving return of spontaneous circulation after resuscitation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-12-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
optic nerve sheath diameter (ONSD) | 7 days
  ONSD measured by ultrasonography during the post-arrest care
carotid artery resistance | 7 days
  carotid artery resistance measured by ultrasonography during the post-arrest care
middle cerebral artery resistance | 7 days
  middle cerebral artery resistance measured by ultrasonography during the post-arrest care

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ching Lien, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No